CLINICAL TRIAL: NCT00209235
Title: Natural History Study of Albright Hereditary Osteodystrophy: Includes Substudies on Effects of Growth Hormone in Patients With Pseudohypoparathyroidism Type 1A and Cognitive & Behavioral Studies in Albright Hereditary Osteodystrophy
Brief Title: Albright Hereditary Osteodystrophy: Natural History, Growth, and Cognitive/Behavioral Assessments
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Connecticut Children's Medical Center (Other)
Collaborators: Johns Hopkins University (Other); Hugo W. Moser Research Institute at Kennedy Krieger, Inc. (Other); UConn Health (Other); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Emily Germain-Lee, Prof of Pediatrics & Prof of Reconstructive Sciences, Director of Albright Center, Head of Academic Affairs & Research, Pediatric Endocrinology, Connecticut Children's Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 16-110; R21HD078864 (NIH)
Record Dates: First submitted 2005-09-13; First posted 2005-09-21 (Estimated); Last update posted 2025-05-28 (Actual); Status verified 2025-05

CONDITIONS: Pseudohypoparathyroidism Type 1A; Albright Hereditary Osteodystrophy; Pseudopseudohypoparathyroidism
Keywords: Pseudohypoparathyroidism Type 1A (PHP 1A); Albright Hereditary Osteodystrophy (AHO); Pseudopseudohypoparathyroidism (PPHP); Growth Hormone Deficiency; Cognition and Behavior
MeSH Terms: conditions — Pseudohypoparathyroidism; Pseudopseudohypoparathyroidism; Dwarfism, Pituitary; Behavior

STUDY DESIGN:
Intervention Model Description: Natural history
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- AHO:neurocognitive and pyschosocial (Experimental): Neurocognitive and psychosocial testing
  Interventions: Behavioral: Neurocognitive and psychosocial testing

INTERVENTIONS:
Behavioral: Neurocognitive and psychosocial testing — Neurocognitive and psychosocial testing

SUMMARY:
We, the researchers, are following the natural history of Albright hereditary osteodystrophy. We have found that growth hormone deficiency is very common in patients with pseudohypoparathyroidism type 1A, which falls under the broader condition termed Albright hereditary osteodystrophy. Patients with pseudohypoparathyroidism type 1A typically are short and obese. Some of these patients are not short during childhood, but due to a combination of factors, they end up short as adults. We are evaluating the effect of growth hormone treatment in those patients with pseudohypoparathyroidism type 1A who are found to be growth hormone deficient (under R01 FD002568, IND 67148, which ended); those who are growth hormone sufficient and were found to have a positive clinical response to growth hormone in a prior clinical trial (under R01 FD00FD003409, IND 67148, which ended); or those who meet the criteria of idiopathic short stature or SGA.

We are also evaluating neurocognitive and psychosocial functioning in participants with AHO in order to determine the specific impairments that are most common in the condition and to determine the best approach toward management.

Funding source -- Growth hormone study: FDA OOPD [R01 FD003409 (which has ended) and R01 FD002568 (which has ended)] Cognitive/behavior: NICHD R21 HD078864 (which has ended)

DETAILED DESCRIPTION:
Pseudohypoparathyroidism type 1A (PHP1A) is a disorder that causes many endocrine and developmental problems. To date, medical treatment has focused primarily on maintenance of normal serum levels of calcium, phosphorous, and thyroid hormone. However, these therapeutic interventions do not address the problems of short stature, obesity, and subcutaneous ossifications, which for many are a source of considerable morbidity and personal distress. These patients require frequent medical care, blood tests, and medication adjustments. PHP1A is an inherited condition with an estimated prevalence in the United States of 1:15,000- 20,000, and the studies that we propose provide an opportunity to improve the quality of life in affected patients. We have found that growth hormone (GH) deficiency is common in these patients, and our data suggest that GH testing should be part of their routine standard of care. We are investigating whether GH treatment can increase final adult height. We are also investigating whether GH treatment can reduce weight and improve a variety of metabolic disturbances and overall health in both children and adults.

GH deficiency not only leads to short stature and obesity, but also to osteoporosis, hyperlipidemia, depressed cardiac and renal function, as well as an overall lack of energy. It is quite possible that treatment of GH-deficient patients with PHP1A could improve any or all of the above problems. GH treatment has been FDA approved for use in both children and adults with GH deficiency. Therefore, it may be possible to provide improvement in health and overall quality of life in these patients.

Additionally, we completed a study in which we treated children with PHP1A who are not GH deficient (i.e., GH sufficient). The rationale is that GH treatment could maximize linear growth velocity prior to the premature bone fusion that occurs in this condition and potentially improve final adult height. The supply of growth hormone has ended for this study, and we are following those participants who were in this study and received the growth hormone supply. Some of these patients remain on growth hormone as per clinical care secondary to their responses.

This study also seeks to define the specific neurocognitive and psychosocial disabilities in individuals with AHO in order to develop therapies and improve quality of life. AHO includes two subtypes: pseudohypoparathyroidism type 1A (PHP1A) and pseudopseudohypoparathyroidism (PPHP).

ELIGIBILITY:
Inclusion Criteria for GH study:

* Diagnosis of pseudohypoparathyroidism type 1A with mutation confirmation
* For the portion of the study in which growth hormone is used for participants who are not growth hormone deficient (ie., growth hormone sufficient), the participant must be over 3 years of age (ie., after 3rd birthday) AND also be pre-pubertal at the time of GH initiation.
* As of now, the growth hormone sufficient participants must meet the FDA-approved criteria for idiopathic short stature or the SGA indication.

Therefore, for all participants enrolling in the growth hormone portion of this study as of now, the growth hormone is used according to FDA-approved indications, and growth hormone use is according to standard of care clinical guidelines.

Exclusion:

* Absence of above diagnosis and failure to meet above criteria

Inclusion Criteria for cognitive/behavioral studies:

* Confirmed diagnosis of Pseudohypoparathyroidism type 1A and Pseudopseudohypoparathyroidism with mutation confirmation
* Ages 4 - 65 yrs

Exclusion:

* Absence of above

Inclusion Criteria for Natural History Study:

* Confirmed diagnosis of Pseudohypoparathyroidism type 1A or Pseudopseudohypoparathyroidism with mutation confirmation
* Ages 0.2 yrs - 89 yrs

Exclusion:

* Absence of above

Ages: 2 Months to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2003-01; Primary Completion 2030-10 (Estimated); Study Completion 2030-12 (Estimated)

PRIMARY OUTCOMES:
PHP1A: Effect of GH on height, growth velocity, final height in children. Effect on weight, BMI, lipids, BMD, self-esteem in all ages. | until achieve final height (approximately 12-15 years)
  Effect of growth hormone
Cognitive and behavioral function in Albright hereditary osteodystrophy | participant will be assessed on day 1; assessment may extend into day 2
  Cognitive and behavioral function assessments/questionnaires

CONTACTS AND LOCATIONS:
Overall Officials: Emily L Germain-Lee, MD, Principal Investigator — Connecticut Children's Medical Ctr. and Univ. of Connecticut School of Medicine
Locations (1):
- Connecticut Children's Medical Center, Hartford, Connecticut, United States

REFERENCES:
- [Background] Germain-Lee EL, Groman J, Crane JL, Jan de Beur SM, Levine MA. Growth hormone deficiency in pseudohypoparathyroidism type 1a: another manifestation of multihormone resistance. J Clin Endocrinol Metab. 2003 Sep;88(9):4059-69. doi: 10.1210/jc.2003-030028. PMID 12970262
- [Background] Germain-Lee EL, Ding CL, Deng Z, Crane JL, Saji M, Ringel MD, Levine MA. Paternal imprinting of Galpha(s) in the human thyroid as the basis of TSH resistance in pseudohypoparathyroidism type 1a. Biochem Biophys Res Commun. 2002 Aug 9;296(1):67-72. doi: 10.1016/s0006-291x(02)00833-1. PMID 12147228
- [Background] Germain-Lee EL, Schwindinger W, Crane JL, Zewdu R, Zweifel LS, Wand G, Huso DL, Saji M, Ringel MD, Levine MA. A mouse model of albright hereditary osteodystrophy generated by targeted disruption of exon 1 of the Gnas gene. Endocrinology. 2005 Nov;146(11):4697-709. doi: 10.1210/en.2005-0681. Epub 2005 Aug 11. PMID 16099856
- [Background] Levine MA, Germain-Lee E, Jan de Beur S. Genetic basis for resistance to parathyroid hormone. Horm Res. 2003;60 Suppl 3:87-95. doi: 10.1159/000074508. PMID 14671404
- [Background] Jan de Beur S, Ding C, Germain-Lee E, Cho J, Maret A, Levine MA. Discordance between genetic and epigenetic defects in pseudohypoparathyroidism type 1b revealed by inconsistent loss of maternal imprinting at GNAS1. Am J Hum Genet. 2003 Aug;73(2):314-22. doi: 10.1086/377136. Epub 2003 Jul 11. PMID 12858292
- [Background] Huso DL, Edie S, Levine MA, Schwindinger W, Wang Y, Juppner H, Germain-Lee EL. Heterotopic ossifications in a mouse model of albright hereditary osteodystrophy. PLoS One. 2011;6(6):e21755. doi: 10.1371/journal.pone.0021755. Epub 2011 Jun 29. PMID 21747923
- [Background] Myllyla RM, Haapasaari KM, Palatsi R, Germain-Lee EL, Hagg PM, Ignatius J, Tuukkanen J. Multiple miliary osteoma cutis is a distinct disease entity: four case reports and review of the literature. Br J Dermatol. 2011 Mar;164(3):544-52. doi: 10.1111/j.1365-2133.2010.10121.x. Epub 2011 Feb 17. PMID 21062265
- [Background] Mantovani G, Bastepe M, Monk D, de Sanctis L, Thiele S, Usardi A, Ahmed SF, Bufo R, Choplin T, De Filippo G, Devernois G, Eggermann T, Elli FM, Freson K, Garcia Ramirez A, Germain-Lee EL, Groussin L, Hamdy N, Hanna P, Hiort O, Juppner H, Kamenicky P, Knight N, Kottler ML, Le Norcy E, Lecumberri B, Levine MA, Makitie O, Martin R, Martos-Moreno GA, Minagawa M, Murray P, Pereda A, Pignolo R, Rejnmark L, Rodado R, Rothenbuhler A, Saraff V, Shoemaker AH, Shore EM, Silve C, Turan S, Woods P, Zillikens MC, Perez de Nanclares G, Linglart A. Diagnosis and management of pseudohypoparathyroidism and related disorders: first international Consensus Statement. Nat Rev Endocrinol. 2018 Aug;14(8):476-500. doi: 10.1038/s41574-018-0042-0. PMID 29959430
- [Background] Mantovani G, Bastepe M, Monk D, de Sanctis L, Thiele S, Ahmed SF, Bufo R, Choplin T, De Filippo G, Devernois G, Eggermann T, Elli FM, Garcia Ramirez A, Germain-Lee EL, Groussin L, Hamdy NAT, Hanna P, Hiort O, Juppner H, Kamenicky P, Knight N, Le Norcy E, Lecumberri B, Levine MA, Makitie O, Martin R, Martos-Moreno GA, Minagawa M, Murray P, Pereda A, Pignolo R, Rejnmark L, Rodado R, Rothenbuhler A, Saraff V, Shoemaker AH, Shore EM, Silve C, Turan S, Woods P, Zillikens MC, Perez de Nanclares G, Linglart A. Recommendations for Diagnosis and Treatment of Pseudohypoparathyroidism and Related Disorders: An Updated Practical Tool for Physicians and Patients. Horm Res Paediatr. 2020;93(3):182-196. doi: 10.1159/000508985. Epub 2020 Aug 5. PMID 32756064
- [Background] Crane JL, Shamblott MJ, Axelman J, Hsu S, Levine MA, Germain-Lee EL. Imprinting status of Galpha(s), NESP55, and XLalphas in cell cultures derived from human embryonic germ cells: GNAS imprinting in human embryonic germ cells. Clin Transl Sci. 2009 Oct;2(5):355-60. doi: 10.1111/j.1752-8062.2009.00148.x. PMID 20443919
- [Result] Germain-Lee EL. Short stature, obesity, and growth hormone deficiency in pseudohypoparathyroidism type 1a. Pediatr Endocrinol Rev. 2006 Apr;3 Suppl 2:318-27. PMID 16675931
- [Result] Long DN, McGuire S, Levine MA, Weinstein LS, Germain-Lee EL. Body mass index differences in pseudohypoparathyroidism type 1a versus pseudopseudohypoparathyroidism may implicate paternal imprinting of Galpha(s) in the development of human obesity. J Clin Endocrinol Metab. 2007 Mar;92(3):1073-9. doi: 10.1210/jc.2006-1497. Epub 2006 Dec 12. PMID 17164301
- [Result] Hsu SC, Groman JD, Merlo CA, Naughton K, Zeitlin PL, Germain-Lee EL, Boyle MP, Cutting GR. Patients with mutations in Gsalpha have reduced activation of a downstream target in epithelial tissues due to haploinsufficiency. J Clin Endocrinol Metab. 2007 Oct;92(10):3941-8. doi: 10.1210/jc.2007-0271. Epub 2007 Jul 24. PMID 17652219
- [Result] Plagge A, Kelsey G, Germain-Lee EL. Physiological functions of the imprinted Gnas locus and its protein variants Galpha(s) and XLalpha(s) in human and mouse. J Endocrinol. 2008 Feb;196(2):193-214. doi: 10.1677/JOE-07-0544. PMID 18252944
- [Result] Long DN, Levine MA, Germain-Lee EL. Bone mineral density in pseudohypoparathyroidism type 1a. J Clin Endocrinol Metab. 2010 Sep;95(9):4465-75. doi: 10.1210/jc.2010-0498. Epub 2010 Jul 7. PMID 20610593
- [Result] Joseph AW, Shoemaker AH, Germain-Lee EL. Increased prevalence of carpal tunnel syndrome in albright hereditary osteodystrophy. J Clin Endocrinol Metab. 2011 Jul;96(7):2065-73. doi: 10.1210/jc.2011-0013. Epub 2011 Apr 27. PMID 21525160
- [Result] Muniyappa R, Warren MA, Zhao X, Aney SC, Courville AB, Chen KY, Brychta RJ, Germain-Lee EL, Weinstein LS, Skarulis MC. Reduced insulin sensitivity in adults with pseudohypoparathyroidism type 1a. J Clin Endocrinol Metab. 2013 Nov;98(11):E1796-801. doi: 10.1210/jc.2013-1594. Epub 2013 Sep 12. PMID 24030943
- [Result] Lin MH, Numbenjapon N, Germain-Lee EL, Pitukcheewanont P. Progressive osseous heteroplasia, as an isolated entity or overlapping with Albright hereditary osteodystrophy. J Pediatr Endocrinol Metab. 2015 Jul;28(7-8):911-8. doi: 10.1515/jpem-2014-0435. PMID 25894639
- [Result] Salemi P, Skalamera Olson JM, Dickson LE, Germain-Lee EL. Ossifications in Albright Hereditary Osteodystrophy: Role of Genotype, Inheritance, Sex, Age, Hormonal Status, and BMI. J Clin Endocrinol Metab. 2018 Jan 1;103(1):158-168. doi: 10.1210/jc.2017-00860. PMID 29059381
- [Result] Germain-Lee EL. Management of pseudohypoparathyroidism. Curr Opin Pediatr. 2019 Aug;31(4):537-549. doi: 10.1097/MOP.0000000000000783. PMID 31145125
- [Result] McMullan P, Maye P, Yang Q, Rowe DW, Germain-Lee EL. Parental Origin of Gsalpha Inactivation Differentially Affects Bone Remodeling in a Mouse Model of Albright Hereditary Osteodystrophy. JBMR Plus. 2021 Nov 16;6(1):e10570. doi: 10.1002/jbm4.10570. eCollection 2022 Jan. PMID 35079678
- [Result] McMullan P, Germain-Lee EL. Aberrant Bone Regulation in Albright Hereditary Osteodystrophy dueto Gnas Inactivation: Mechanisms and Translational Implications. Curr Osteoporos Rep. 2022 Feb;20(1):78-89. doi: 10.1007/s11914-022-00719-w. Epub 2022 Feb 28. PMID 35226254
- [Result] Krishnan N, McMullan P, Yang Q, Buscarello AN, Germain-Lee EL. Prevalence of Chiari malformation type 1 is increased in pseudohypoparathyroidism type 1A and associated with aberrant bone development. PLoS One. 2023 Jan 20;18(1):e0280463. doi: 10.1371/journal.pone.0280463. eCollection 2023. PMID 36662765
- See also: website for Dr. Germain-Lee's clinical trials and research — https://www.connecticutchildrens.org/about-us/find-a-doctor/emily-l-germain-lee-md/
- See also: website for Dr. Germain-Lee's UConn Health profile — http://facultydirectory.uchc.edu/profile?profileId=Germain-Lee-Emily